CLINICAL TRIAL: NCT05762042
Title: Comparison of the Efficacy and Tolerability of Femal Versus Placebo in the Treatment of Hot Flashes in Patients With Previous Breast Cancer
Brief Title: Comparison of the Efficacy and Tolerability of Femal Versus Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Ordine Mauriziano di Torino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FEMAL
Record Dates: First submitted 2023-02-16; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Menopause
MeSH Terms: conditions — Breast Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femal (Experimental): Patients in this arm will receive FEMAL (2 cp/die) for three months long
  Interventions: Other: dietary supplement
- Placebo (Placebo Comparator): Patients in this arm will receive PLACEBO (2 cp/die) for three months long
  Interventions: Other: dietary supplement

INTERVENTIONS:
Other: dietary supplement — Femal, a food supplement based on pollen extracts introduced in Europe in 1999, is a non-estrogenic alternative to hormone replacement therapy in women with vasomotor symptoms.
  The mechanism of action of Femal has not yet been fully clarified: Femal inhibits the absorption of serotonin in a dose-dependent manner and has strong antioxidant properties.
  The lack of estrogenic effects would make this preparation of particular interest for women with a previous hormone-dependent neoplasia who undergo an early iatrogenic menopause.
  Femal tablets contain a standardized formulation containing: GC Fem pollen extract 40 mg, PI82 pollen / pistil extract 120 mg, vitamin E 5 mg, amino acids 14 mg per tablet.
  The dosage is 2 tablets a day orally.

SUMMARY:
Femal, a food supplement based on pollen extracts introduced in Europe in 1999, is a non-estrogenic alternative to hormone replacement therapy in women with vasomotor symptoms.

Patients with prior breast cancer, spontaneous or iatrogenic menopause or who are premenopausal with ovarian function suppressed by GNRH analogue and experiencing severe vasomotor symptoms (at least 20 hot flashes per week) will be included.

Patients who are on tamoxifen or anti-estrogen or aromatase inhibitor therapy are eligible if started at least 2 months prior to study entry.

Patients on SSRI or SNRI antidepressant therapy are excluded. Eligible patients will be randomly assigned to either Femal (2 cp/day) or placebo (2 cp/day) for 3 months (double-blind study).

ELIGIBILITY:
Inclusion Criteria:

- patients with a history of breast cancer, in spontaneous or iatrogenic menopause or who are premenopausal with ovarian function suppressed by GNRH analogue and experiencing severe vasomotor symptoms (at least 20 hot flushes per week).

Patients who are on tamoxifen or aromatase anti-estrogen or aromatase inhibitor therapy are eligible if started at least 2 months prior to study entry

Exclusion Criteria:

* Patients on SSRI or SNRI antidepressant therapy are excluded

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
efficacy of Femal in reducing the mean score of vasomotor symptoms between baseline (T0) and month 3 (T2). | 3 months
  verify efficacy of Femal in reducing the mean score of vasomotor symptoms between baseline (T0) and month 3 (T2).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Europeo di Oncologia, Milan
  - Policlinico Gemelli di Roma, Roma